CLINICAL TRIAL: NCT07201298
Title: A Prospective Contralateral Comparison of Ray-Tracing Guided LASIK (WaveLight® Plus LASIK) vs. Small Incision Lenticule Extraction (SMILE® Pro) Using VisuMax® 800, or Wavefront Optimized LASIK or Topography Guided LASIK (Contoura LASIK): A Three-Phase Visual Outcomes Study.
Brief Title: A Three-Phase Contralateral Comparison of Ray-Tracing Guided LASIK Versus Three Other Refractive Surgery Platforms to Correct Myopia or Myopia With Astigmatism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hoopes Vision (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMRC-WLP-VWC
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Myopia; Astigmatism
Keywords: refractive surgery; myopia; astigmatism; excimer laser; femtosecond laser; Ray Tracing; Lenticule; SMILE; KLEx; Contoura; Topography Guided LASIK; Wavefront Optimized
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Intervention Model Description: A= Ray-Tracing Guided LASIK (RTGL) B= Keratorefractive Lenticule Extraction (KLEx) C=WaveFront Optimized LASIK (WFOL) D= Topography Guided LASIK (TGL)
  This is a contralateral eye study with 3 different phases:
  Phase 1 has 2 Arms: Arm 1 consists of 22 subjects who have RTGL in the Right Eye and KLEx in the Left Eye, Arm 2 consists of 22 subjects who have KLEx in the Right Eye and RTGL in the Left Eye.
  Phase 2 has 2 Arms: Arm 1 consists of 22 subjects who have RTGL in the Right Eye and WFOL in the Left Eye, Arm 2 consists of 22 subjects who have WFOL in the Right Eye and RTGL in the Left Eye.
  Phase 3 has 2 Arms: Arm 1 consists of 22 subjects who have RTGL in the Right Eye and TGL in the Left Eye, Arm 2 consists of 22 subjects who have TGL in the Right Eye and RTGL in the Left Eye.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (6):
- ARM 1: Ray Tracing Guided LASIK in OD and Keratorefractive Lenticule Extraction in OS (Active Comparator): Subjects receive Ray Tracing Guided LASIK in the RIGHT EYE and Keratorefractive Lenticule Extraction in the LEFT EYE
  Interventions: Device: Ray-Tracing Guided LASIK; Device: Keratorefractive Lenticule Extraction (KLEx)
- ARM 2: WaveLight Plus LASIK in OS and Keratorefractive Lenticule Extraction in OD (Active Comparator): Subjects receive Ray Tracing Guided LASIK in the LEFT EYE and Keratorefractive Lenticule Extraction in the RIGHT EYE
  Interventions: Device: Ray-Tracing Guided LASIK; Device: Keratorefractive Lenticule Extraction (KLEx)
- ARM 3: Ray Tracing Guided LASIK in OD and Wavefront Optimized LASIK in OS (Active Comparator): Subjects receive Ray Tracing Guided LASIK in the RIGHT EYE and Wavefront Optimized LASIK in the LEFT EYE.
  Interventions: Device: Ray-Tracing Guided LASIK; Device: WaveFront Optimized LASIK
- ARM 4: Ray Tracing Guided LASIK in OS and Wavefront Optimized LASIK in OD (Active Comparator): Subjects receive Ray Tracing Guided LASIK in the LEFT EYE and Wavefront Optimized LASIK in the RIGHT EYE
  Interventions: Device: Ray-Tracing Guided LASIK; Device: WaveFront Optimized LASIK
- ARM 5: Ray Tracing Guided LASIK in OD and Topography Guided LASIK in OS (Active Comparator): Subjects receive Ray Tracing Guided in the RIGHT EYE and Topography Guided LASIK in the LEFT EYE
  Interventions: Device: Ray-Tracing Guided LASIK; Device: Topography Guided LASIK
- ARM 6: Ray Tracing Guided LASIK in OS and Topography Guided LASIK in OD (Active Comparator): Subjects receive Ray Tracing Guided LASIK in the LEFT EYE and Topography Guided LASIK in the RIGHT EYE
  Interventions: Device: Ray-Tracing Guided LASIK; Device: Topography Guided LASIK

INTERVENTIONS:
Device: Ray-Tracing Guided LASIK — A form of LASIK where Ray-Tracing technology is used to create the surgical profile for treating the cornea.
Device: Keratorefractive Lenticule Extraction (KLEx) — A form of corneal refractive surgery utilizing a femtosecond laser to create a lens shaped lenticule of corneal tissue that is removed through a small corneal incision.
  Arms: ARM 1: Ray Tracing Guided LASIK in OD and Keratorefractive Lenticule Extraction in OS; ARM 2: WaveLight Plus LASIK in OS and Keratorefractive Lenticule Extraction in OD
Device: WaveFront Optimized LASIK — A form of LASIK where the corneal treatment profile is modified to decrease induced Spherical Aberration.
  Arms: ARM 3: Ray Tracing Guided LASIK in OD and Wavefront Optimized LASIK in OS; ARM 4: Ray Tracing Guided LASIK in OS and Wavefront Optimized LASIK in OD
Device: Topography Guided LASIK — A form of LASIK where a corneal topography of the cornea is used to create the surgical profile for treating the cornea.
  Arms: ARM 5: Ray Tracing Guided LASIK in OD and Topography Guided LASIK in OS; ARM 6: Ray Tracing Guided LASIK in OS and Topography Guided LASIK in OD

SUMMARY:
This purpose of this study is to compare a new form of LASIK called Ray Tracing Guided LASIK to 3 other forms of corneal refractive surgery: 1. KLEx (KeratoLenticule Extraction) using the Zeiss Visumax 800 Laser, 2. WFO LASIK (Wavefront Optimized LASIK) using the Alcon EX500 Laser, and 3. Topography Guided LASIK (Contoura LASIK) also using the Alcon EX500 Laser.

DETAILED DESCRIPTION:
This is a prospective, randomized, simultaneous, contralateral eye study comparing visual outcomes for 4 different refractive technologies. This study will be conducted in 3 phases. Each phase will include at least 44 subjects undergoing refractive correction surgery for myopia or myopia with astigmatism. Each phase will compare Ray-Tracing LASIK to 1 of 3 other forms of corneal refractive surgery. The Phase 1 comparator will be KLEx (KeratoLenticule Extraction) using the Zeiss Visumax 800 Laser. The Phase 2 comparator will be WFO LASIK (Wavefront Optimized LASIK) using the Alcon EX500 Laser. The Phase 3 comparator will be Topography Guided LASIK (Contoura LASIK) also using the Alcon EX500 Laser. Patients will be selected from the Hoopes Vision patient population after a preliminary refractive evaluation has been completed. Patients who express an interest in the study will be consented. After informed consent has been obtained and the patient has completed a screening exam and met all study criteria they will be considered enrolled. For each Phase, randomization will ensure 50% of Right Eyes will receive Ray-Tracing LASIK and 50% of Right Eyes will receive the other comparator procedure. Subjects will be given postoperative care instructions and medications following standard of care practices. Subjects will return for a 1-day, 1-week, 1-month, 3-month, 6-month, and 12-month visit. Retreatments may only occur after all postoperative study visits have been completed and/or the subject has exited the study. At the preliminary screening visit, 1-month, 3-month, 6-month and 12-mont postoperative visits, patients will complete a Patient Participant Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Age 22-50 at the time of consent
2. Diagnosis of myopia or myopia with astigmatism with Preoperative manifest spherical equivalent refraction of ≥ -2.00 and ≤ -9.00 D (-2.00 D through -9.00 D)
3. Preop Spherical component of ≥ -2.00 and ≤ -8.00 D (-2.00 D through -8.00 D)
4. Refractive Cylinder of ≤ -3.00 D (0.00 through -3.00 D)
5. BCVA of 20/20 or better in each eye (83 or more letters on the ETDRS Chart)
6. Subjects must have a stable refraction which is defined as a change in spherical equivalent no greater than 0.50 D comparing the screening visit manifest refraction to a previous refraction, spectacle Rx, or contact lens Rx, 12 months or older.
7. Subjects who are contact lens wearers must discontinue the use of soft lenses (spherical or toric) for at least 5 days and hard or gas-permeable lenses for at least 4 weeks prior to the preoperative screening evaluation. Hard or gas-permeable lens wearers must not return to contact lens use before surgery. Soft lens wearers may resume contact lens wear after all preoperative testing is completed, but must discontinue lens use at least 5 days before surgery.
8. Acceptable preoperative tomography and examination results for refractive procedures as determined by the Principal Investigator.
9. Surgical plan includes treatment target for emmetropia in both eyes, and no monovision.
10. Subject is capable and willing to use postoperative medications as prescribed.
11. Subject has ability to successfully complete all preoperative and postoperative questionnaires, testing, and exam visits.
12. Subject is willing and able to return for all postoperative examinations.

Exclusion Criteria:

1. Clinically significant dry eye on clinical examination, as determined by the investigator
2. Irregular astigmatism, keratoconus, keratoconus suspect, or abnormal corneal tomography
3. History of corneal dystrophies or guttata
4. History of herpetic keratitis or active disease
5. History of prior refractive surgery
6. History of glaucoma or glaucoma suspect
7. History of uncontrolled diabetes, unstable hypertension, or unstable autoimmune disease.
8. Females who are pregnant, breastfeeding, or intend to become pregnant any time during the study as determined by verbal inquiry.
9. The Principal Investigator has determined the subject not to be a good candidate for the study.

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Uncorrected Visual Acuity | 3, 6 and 12 month
  Percentage of eyes acheiving uncorrected visual acuity of 20/40, 20/25, 20/20, 20/16, 20/12.5, and 20/10 at post-operative month 3, 6 and 12

SECONDARY OUTCOMES:
Predictability | 3, 6, and 12 months
  Percentage of eyes that acheive MRSE within +/- 0.5 diopters and +/- 1.00 diopters of intended correction at post-operative visits 3, 6, and 12-months.

CONTACTS AND LOCATIONS:
Overall Officials: Majid Moshirfar, MD, Principal Investigator — Hoopes Vision
Locations (1):
- Hoopes Moshirfar Research Center, Draper, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Khoramnia R, Lohmann CP, Wuellner C, Kobuch KA, Donitzky C, Winkler von Mohrenfels C. Effect of 3 excimer laser ablation frequencies (200 Hz, 500 Hz, 1000 Hz) on the cornea using a 1000 Hz scanning-spot excimer laser. J Cataract Refract Surg. 2010 Aug;36(8):1385-91. doi: 10.1016/j.jcrs.2010.01.033. PMID 20656164
- [Background] Winkler von Mohrenfels C, Khoramnia R, Lohmann CP. Comparison of different excimer laser ablation frequencies (50, 200, and 500 Hz). Graefes Arch Clin Exp Ophthalmol. 2009 Nov;247(11):1539-45. doi: 10.1007/s00417-009-1102-x. Epub 2009 Jul 14. PMID 19597838
- [Background] Meidani A, Tzavara C. Comparison of efficacy, safety, and predictability of laser in situ keratomileusis using two laser suites. Clin Ophthalmol. 2016 Aug 24;10:1639-46. doi: 10.2147/OPTH.S110626. eCollection 2016. PMID 27601880
- [Background] Mrochen M, Donitzky C, Wullner C, Loffler J. Wavefront-optimized ablation profiles: theoretical background. J Cataract Refract Surg. 2004 Apr;30(4):775-85. doi: 10.1016/j.jcrs.2004.01.026. PMID 15093638
- [Background] Mrochen M, Seiler T. Influence of corneal curvature on calculation of ablation patterns used in photorefractive laser surgery. J Refract Surg. 2001 Sep-Oct;17(5):S584-7. doi: 10.3928/1081-597X-20010901-15. PMID 11583235
- [Background] Ganesh S, Brar S, Swamy DT. Comparison of Clinical Outcomes and Patient Satisfaction Following SMILE Performed With the VisuMax 800 in One Eye and VisuMax 500 in the Contralateral Eye. J Refract Surg. 2025 Jan;41(1):e14-e21. doi: 10.3928/1081597X-20241113-02. Epub 2025 Jan 1. PMID 39783817
- [Background] Reinstein DZ, Archer TJ, Potter JG, Gupta R, Wiltfang R. Refractive and Visual Outcomes of SMILE for Compound Myopic Astigmatism With the VISUMAX 800. J Refract Surg. 2023 May;39(5):294-301. doi: 10.3928/1081597X-20230301-02. Epub 2023 May 1. PMID 37162399
- [Background] Teus MA, Garcia-Gonzalez M. Comparison of the visual results after small incision lenticule extraction and femtosecond laser-assisted LASIK for myopia. J Refract Surg. 2014 Sep;30(9):582. doi: 10.3928/1081597X-20140819-01. No abstract available. PMID 25208349
- [Background] Pinero DP, Teus MA. Clinical outcomes of small-incision lenticule extraction and femtosecond laser-assisted wavefront-guided laser in situ keratomileusis. J Cataract Refract Surg. 2016 Jul;42(7):1078-93. doi: 10.1016/j.jcrs.2016.05.004. PMID 27492109
- [Background] Ganesh S, Gupta R. Comparison of visual and refractive outcomes following femtosecond laser- assisted lasik with smile in patients with myopia or myopic astigmatism. J Refract Surg. 2014 Sep;30(9):590-6. doi: 10.3928/1081597X-20140814-02. PMID 25250415
- [Background] Shah R, Shah S, Sengupta S. Results of small incision lenticule extraction: All-in-one femtosecond laser refractive surgery. J Cataract Refract Surg. 2011 Jan;37(1):127-37. doi: 10.1016/j.jcrs.2010.07.033. PMID 21183108
- [Background] Sekundo W, Kunert KS, Blum M. Small incision corneal refractive surgery using the small incision lenticule extraction (SMILE) procedure for the correction of myopia and myopic astigmatism: results of a 6 month prospective study. Br J Ophthalmol. 2011 Mar;95(3):335-9. doi: 10.1136/bjo.2009.174284. Epub 2010 Jul 3. PMID 20601657
- [Background] Blum M, Taubig K, Gruhn C, Sekundo W, Kunert KS. Five-year results of Small Incision Lenticule Extraction (ReLEx SMILE). Br J Ophthalmol. 2016 Sep;100(9):1192-5. doi: 10.1136/bjophthalmol-2015-306822. Epub 2016 Jan 8. PMID 26746577
- [Background] Reinstein DZ, Archer TJ, Gobbe M. Small incision lenticule extraction (SMILE) history, fundamentals of a new refractive surgery technique and clinical outcomes. Eye Vis (Lond). 2014 Oct 16;1:3. doi: 10.1186/s40662-014-0003-1. eCollection 2014. PMID 26605350
- [Background] Lee JK, Chuck RS, Park CY. Femtosecond laser refractive surgery: small-incision lenticule extraction vs. femtosecond laser-assisted LASIK. Curr Opin Ophthalmol. 2015 Jul;26(4):260-4. doi: 10.1097/ICU.0000000000000158. PMID 26058022